CLINICAL TRIAL: NCT00000299
Title: Rapid Opiate Detoxification & Naltrexone Induction Using Bup.
Brief Title: Rapid Opiate Detoxification and Naltrexone Induction Using Buprenorphine - 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Walter Ling, PI, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NIDA-09260-2; P50DA009260 (NIH); P50-09260-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Opioid-Related Disorders
Keywords: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- buprenorphine (Active Comparator): depot buprenorphine
  Interventions: Drug: Buprenorphine
- buprenorphine and ultra-low dose naloxone (Experimental): depot buprenorphine and naloxone
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to develop a clinical protocol to detoxify patients from opiates to naltrexone using buprenorphine and to develop pilot data for a grant application for a controlled study of the efficacy of the new clinical protocol for outpatients.

ELIGIBILITY:
Inclusion Criteria:

Males/Females, ages 21-50. Opiate dependence according to DSM-IV criteria. Self-reported use within the last 30 days. Agreeable to conditions of study and signed informed consent.

Exclusion Criteria:

psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nursing women. Dependent on etoh or benzodiazepines or other sedative-hypnotics. Acute hepatitis. Other medical conditions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Opiate craving | 10 test days
  opiate craving is measured on each test day.
Opiate withdrawal symptoms | 10 test days
  opiate withdrawal symptoms are documented for each test day

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States